CLINICAL TRIAL: NCT03332602
Title: The Effect of Encapsulation Material and Encapsulated Micronutrients on Iron Absorption in Iron Depleted Women Consuming Iron Fortified Bread.
Brief Title: Iron Absorption From Encapsulated Iron Sulphate in Microspheres
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Omnifortificant
Record Dates: First submitted 2017-10-18; First posted 2017-11-06 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Iron-deficiency
Keywords: Iron deficiency; Iron fortification; Iron encapsulation
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- free FeSO4 (Experimental): wheat bread fortified with free FeSO4
  Interventions: Dietary Supplement: free FeSO4
- free FeSO4 and empty microspheres (Experimental): wheat bread fortified with free FeSO4, and empty microspheres
  Interventions: Dietary Supplement: free FeSO4 and empty microspheres
- free FeSO4 with eudragit polymer (Experimental): wheat bread fortified with free FeSO4, and eudragit polymer
  Interventions: Dietary Supplement: free FeSO4 and eudragit polymer
- free FeSO4 with Hyaluronic Acid (Experimental): wheat bread fortified with free FeSO4, and hyaluronic acid
  Interventions: Dietary Supplement: free FeSO4 and hylauronic acid
- encapsulated FeSO4 3.2% (Experimental): wheat bread fortified with encapsulated FeSO4 in a microsphere with 3.2% Fe loading
  Interventions: Dietary Supplement: encapsulated FeSO4 3.2%
- encapsulated FeSO4 20% (Experimental): wheat bread fortified with encapsulated FeSO4 in a microsphere with 20% Fe loading
  Interventions: Dietary Supplement: encapsulated FeSO4 20%
- encapsulated FeSO4 3.2%, encap. Vitamin A (Experimental): wheat bread fortified with encapsulated FeSO4 in a microsphere with 3.2% Fe loading, and encapsulated Vitamin A as microspheres
  Interventions: Dietary Supplement: encapsulated FeSO4 3.2%, encapsulated Vitamin A
- encapsulated FeSO4 3.2%, encap. Vitamin A, free folicacid (Experimental): wheat bread fortified with encapsulated FeSO4 as microsphere with 3.2% Fe loading, encapsulated Vitamin A as microspheres and free folic acid
  Interventions: Dietary Supplement: encapsulated FeSO4 3.2%, encapsulated Vitamin A, free Folic Acid
- FeSO4 embedded in Hyaluronic Acid (Experimental): wheat bread fortified with FeSO4 that is embedded in hyaluronic acid.
  Interventions: Dietary Supplement: FeSO4 embedded in Hyaluronic acid

INTERVENTIONS:
Dietary Supplement: free FeSO4 — Testmeal with free FeSO4
  Arms: free FeSO4
Dietary Supplement: free FeSO4 and empty microspheres — Testmeal with free FeSO4 and empty micropsheres
  Arms: free FeSO4 and empty microspheres
Dietary Supplement: free FeSO4 and hylauronic acid — Testmeal with free FeSO4 and hyaluronic acid
  Arms: free FeSO4 with Hyaluronic Acid
Dietary Supplement: free FeSO4 and eudragit polymer — Testmeal with free FeSO4 and eudragit polymer
  Arms: free FeSO4 with eudragit polymer
Dietary Supplement: encapsulated FeSO4 3.2% — Testmeal with encapsulated FeSO4 with 3.2% Fe loading
  Arms: encapsulated FeSO4 3.2%
Dietary Supplement: encapsulated FeSO4 20% — Testmeal with encapsulated FeSO4 with 20% Fe loading
  Arms: encapsulated FeSO4 20%
Dietary Supplement: encapsulated FeSO4 3.2%, encapsulated Vitamin A — Testmeal with encapsulated FeSO4 with 3.2% Fe loading, and encapsulated Vitamin A
  Arms: encapsulated FeSO4 3.2%, encap. Vitamin A
Dietary Supplement: encapsulated FeSO4 3.2%, encapsulated Vitamin A, free Folic Acid — Testmeal with encapsulated FeSO4 with 3.2% Fe loading, and encapsulated Vitamin A, with free folic acid.
  Arms: encapsulated FeSO4 3.2%, encap. Vitamin A, free folicacid
Dietary Supplement: FeSO4 embedded in Hyaluronic acid — Testmeal with FeSO4 embedded in Hyaluronic acid
  Arms: FeSO4 embedded in Hyaluronic Acid

SUMMARY:
Food fortification has shown to be efficacious to alleviate the burden of micronutrient deficiencies. Ensuring the bioavailability of iron and maintaining the sensory quality and stability of the fortified food and other added micronutrients remains a challenge. Soluble iron compounds cause minor organoleptic changes in foods but their bioavailability in man is rather low. Water-soluble iron compounds, such as ferrous sulphate (FeSO4), are the compounds in which the iron is most bioavailable; however, they often cause unfavorable sensory changes.

Encapsulation of iron has excellent potential for overcoming unwanted sensory changes and iodine losses in salt, while maintaining acceptable bioavailability. In the present project, we would like to investigate the iron bioavailability from a new formulation of encapsulated iron sulphate based on hyaluronic acid (HA) and a polymer from the eudragit family.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 40 years old
* Marginal iron status (PF <25 ng/ml)
* Body weight < 65 kg
* Normal body Mass Index (18.5 - 25 kg/m2)
* Signed informed consent

Exclusion Criteria:

* Pregnancy (assessed by a pregnancy test) / intention to become pregnant
* Lactating up to 6 weeks before study initiation
* Moderate or severe anaemia (Hb < 9.0 g/dL)
* Elevated C reactive Protein (CRP) (> 5.0 mg/L)
* Any metabolic, gastrointestinal kidney or chronic disease such as diabetes, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement)
* Continuous/long-term use of medication during the whole study (except for contraceptives)
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st meal administration
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months
* Earlier participation in a study using Fe stable isotopes or participation in any clinical study within the last 30 days
* Participant who cannot be expected to comply with study protocol (e.g. not available on certain study appointments or difficulties with blood sampling)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the isotopic ratio of iron in blood at week 2 | baseline, 2 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 2 in the isotopic ratio of iron in blood at week 4 | 2 weeks, 4 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 4 in the isotopic ratio of iron in blood at week 6 | 4 weeks, 6 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.

SECONDARY OUTCOMES:
Haemoglobin | baseline, weeks 2, 4 and 6
  Haemoglobin of each timepoint
Plasma Ferritin | baseline, weeks 2, 4 and 6
  Plasma Ferritin of each timepoint
inflammation marker | baseline, weeks 2, 4 and 6
  C reactive Protein of each timepoint

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition Laboratory, ETH Zurich, Zurich, Switzerland